CLINICAL TRIAL: NCT07189039
Title: Studying Access to Healthcare for Children in the Child Welfare System: the Health of Protected Children
Acronym: SESAME
Status: Recruiting | Type: Observational
Sponsor: Fondation Ildys (Other)
Collaborators: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: RI2025_003
Record Dates: First submitted 2025-09-16; First posted 2025-09-23 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Medical Care
Keywords: social services for children; child protection department,; medical care; medical follow-up; medical treatment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Child Protection in France, defined by Article L.112-3 of the Social Action and Family Code (CASF), "aims to ensure that the child's fundamental needs are taken into account, to support his or her physical, emotional, intellectual and social development, and to preserve his or her health, safety, morality and education, while respecting his or her rights". It therefore covers many aspects : prevention, identification of situations of danger or risk of danger, and implementation of administrative or judicial protection measures for minors and adults under 21. This policy is largely entrusted to departmental councils and local authorities with special status, notably through their child welfare services (ASE)" (Reference 1).

According to the report by the National Observatory for Child Protection (ONPE), by the end of 2022, the number of minors in care, all child protection services and measures combined, would be 310,577 minors, while the number of young adults in care would be 34,105 adults (Reference 2). Between 2011 and 2022, the estimated number of minors will increase by 13%, while the estimated number of young adults will rise by 62% (Reference 2).

The assessment of a child's health preservation during a child protection measure is governed by the following texts:

* Code de l'Action Sociale et des Familles (CASF) (Social and Family Action Code), Code Civil (Civil Code) and Code de Justice Pénale des mineurs (Juvenile Criminal Justice Code): these define the grounds and nature of administrative and judicial interventions;
* Code de la Santé Publique (CSP) (Public Health Code): defines compulsory examinations according to the child's age, and the procedures to be followed.

The texts have been reformed in recent years by :

* Law n°2007-293 of March 5, 2007 reforming child protection ;
* Law n°2016-297 of March 14, 2016 on child protection;
* Law n°2022-140 of February 7, 2022, known as the "Taquet" law, on child protection.

In the Defender of Rights' framework decision on child protection (Reference 3), it is stated that "due to their history and particular vulnerability, children in child protection care have specific health needs. Numerous studies have demonstrated the deteriorated state of health of these children, the lack of information on risk factors, family history, the need for psychological care, etc.".

These findings have led to the launch, in addition to legal reforms, of innovative national experiments falling within the scope of Article 51 of the French Social Security Financing Act: "Pégase" and "Santé Protégée", two programs designed to coordinate the care of children in the care of the Children's social welfare.

As stated in its strategic plan (Référence 4), "the ILDYS Foundation's action is part of a public service mission in conjunction with the Finistère Child and Family Department. In the child protection sector, the aim is to respond as closely as possible to the needs of each child, and to guarantee his or her safety through support for parenthood and parental substitution."

DETAILED DESCRIPTION:
Within the ILDYS Foundation, the missions of the Social Pole by delegation of the Finistère Departmental Council are therefore to ensure the Protection, Education, and Maintenance of minors under Article L221-1 of the Code of Social Action and Families modified by Law 2016-297 of March 14, 2016.

Since 1991, the Finistère Departmental Council has been setting general objectives for social intervention within the framework of departmental plans drawn up in consultation with all authorized partners. The evolution of the Pôle's projects is therefore set within the context of these reflections and the priorities that emerge from them, as well as the new laws and recommendations of good professional practice that govern our sector. In this way, the Pôle Social provides support for some 262 children in 14 departments, including the following which will be involved in the study:

The Social Children's Home (Maison d'Enfants à Caractère Social (MECS)), which accommodates 40 minors in 3 educational homes located in Brest métropole Océane for young people aged 3 to 18 :

* Le Foyer de Kertatupage
* Le foyer de Plougastel
* Le Foyer de Pont-Neuf Petits et Pont-Neuf Grands

Diversified Family Investment (Placement Familial Diversifié (PFD)) is located in Brest and Landivisiau, on the premises of the Saint-Vincent Lannouchen EHPAD, and can accommodate children with disabilities in a :

* Placement Familial Social (PFS) with 72 places, including 2 outside the department.
* Placement Familial Guidance Parentale (PFGP) with 15 places The Educational support service for independent living (Service d'Accompagnement Educatif à l'Autonomie (SAEA), which supports 13 young people aged 16 to 21 in shared apartments, studios and Foyer Jeunes Travailleurs (FJT).

These three services were selected for this study because they offer long-term accommodation for minors and adults placed with the ILDYS Foundation.

The challenge for the social department is to respond as closely as possible to the needs of children and their families, in line with the Foundation's institutional project.

Public interest justification As mentioned above, the ILDYS foundation takes in and supports young people (minors or adults) entrusted by the Département within its residential services (homes, foster families, SAEA). This support is provided over a long period, averaging five years. This time scale is significant, and will therefore enable us to assess different aspects of the health of children entrusted by the ASE.

So, through this study, the ILDYS Foundation wishes to measure the response to the "standard" but also specific health needs of the protected children entrusted to the Foundation, before their entry and after their entry into the ILDYS Foundation's current service.

This inventory can then be used to issue recommendations aimed at improving the health monitoring of children entrusted to the Child welfare ( Aide Sociale à l'Enfance) system, and their overall health.

Design of study Research Project Not Involving the Human Person (RNIPH). Cross-sectional, multicenter, retrospective descriptive study. Each child's access to care will be determined at the time of inclusion, from birth, focusing on current recommendations (examinations, check-ups, vaccinations), based on the child's medical record.

Two periods will be distinguished: before and after entry into the current ILDYS Foundation service.

ELIGIBILITY:
Inclusion Criteria:

* Protected child
* Aged over 3 or under 21 at the time of inclusion
* Housed in one the three following ILDYS Foundation faicilities : PFS, MECS, SAEA
* For at least 6 months of continuous at the date of inclusion

Exclusion Criteria:

* Minor whose guardian (parent or ASE official if parent has lost parental authorithy) objects to the study being carried out
* Young adult or minor capable of discernment, objecting to the study being carried out

Ages: 3 Years to 21 Years | Sex: All
Age Groups: Child, Adult
Study Population: Protected children aged over 3 or under 21 at the time of inclusion, and must have been accommodated in one of the Foundation's three facilities (PFS, MECS, or SAEA) for at least 6 months of continuous presence at the time of inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 124 (Estimated)
Dates: Start 2025-09-23 (Actual); Primary Completion 2025-09-25 (Estimated); Study Completion 2025-09-25 (Estimated)

PRIMARY OUTCOMES:
Evaluating access to healthcare for children protected by the Foundation's three departments | From July 2025 to september 2025
  Evaluate access to care, in terms of compliance with recommendations, for protected children since their placement within one of the following three ILDYS Foundation services:
  * PFS : Placement Familial Spécialisé;
  * MECS : Maison d'Enfants à Caractère Social;
  * SAEA : Service d'Accompagnement Educatif à l'Autonomie.
  The judging criterion is compliance (yes/no) with recommendations for each of the following themes assessed over the period of presence in one of the ILDYS Foundation services considered:
  * Vaccinations (one item for each vaccination to be carried out during the period in question)
  * Health check-ups (one item for each check-up to be carried out during the period in question)
  * Compulsory medical examinations, compulsory examinations for neurodevelopmental disorders, compulsory dental examinations (one item for each examination to be carried out in the period concerned)
  * Other optional medical or dental examinations
Evaluating access to healthcare for children protected by the Foundation's three departments | from july 2025 to september 2025
  During data collection, the nurse and/or social worker notes, particularly with regard to the child's age, whether for the item in question (e.g. DTP vaccine), public health recommendations have been applied in accordance with the vaccination and compulsory health check-up schedules. It is also noted whether or not the child was present in the ILDYS Foundation's current department at the expected date of the item's compliance check.

SECONDARY OUTCOMES:
Verify access to certain specialists for protected children | from july 2025 to september 2025
  Verify access to certain specialists, in addition to GPs and maternal and child welfare doctors, since the placement of protected children with the ILDYS Foundation.
  Recording of consultations with health specialists other than GPs and maternal and child welfare doctors in the SILAO computerized file or in the child's health record since his or her arrival at one of the ILDYS Foundation establishments.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation ILDYS, Brest, France

IPD SHARING:
Plan to Share IPD: Undecided